CLINICAL TRIAL: NCT01641601
Title: Randomized Controlled Trial of Prehospital Cervical Ripening With an Outpatient Transcervical Foley Balloon and the Duration of Induction and Maternal Satisfaction
Brief Title: Prehospital Cervical Ripening Before Induction and the Maternal Experience
Acronym: "PRIME"
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate enrollment. Key study personnel transitioned to a different role.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-08620
Record Dates: First submitted 2012-07-03; First posted 2012-07-17 (Estimated); Results first posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-07

CONDITIONS: Labor, Induced; Cervical Ripening
Keywords: Induction of labor; Outpatient cervical ripening

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Management (No Intervention): Patients in the usual management arm will have no pre-hospital cervical ripening and will undergo labor induction according to standard labor induction protocols on an inpatient basis.
- Outpatient transcervical Foley balloon (Experimental): Patients in the experimental group will have a 30 cc transcervical Foley balloon placed in the outpatient setting approximately 12-18 hours prior to their labor induction. Once admitted, they will undergo inpatient labor induction as per usual protocols.
  Interventions: Device: Outpatient transcervical Foley balloon

INTERVENTIONS:
Device: Outpatient transcervical Foley balloon — A 30 cc transcervical Foley balloon will be placed in the outpatient setting prior to labor induction.
  Arms: Outpatient transcervical Foley balloon

SUMMARY:
This is a randomized study evaluating the impact of pre-hospital cervical ripening with a transcervical Foley balloon before labor induction in full-term pregnancies on the length of inpatient labor induction and maternal satisfaction with the labor induction process. The investigators hypothesize that women who receive pre-hospital cervical ripening will have a shorter duration of inpatient labor induction as compared to women without pre-hospital cervical ripening.

DETAILED DESCRIPTION:
Labor induction is a common procedure among pregnant patients at term. This process involves a period of cervical preparation ("ripening") for women who have an "unfavorable" cervical examination at the time labor induction is scheduled. Cervical ripening may take place with pharmacologic or mechanical strategies, which at this time are traditionally administered on an inpatient basis. This process can 24 or more hours, resulting in a lengthy hospitalization with the associated costs and frustrations for both patients and L&D staff.

The proposed study is a randomized, controlled trial to explore the following research question: Among women with full-term pregnancies requiring labor induction, does pre-hospital, outpatient cervical ripening reduce the amount of inpatient time needed to achieve delivery as compared to no pre-hospital cervical ripening? As a secondary objective, we also wish to explore if outpatient cervical ripening is acceptable to patients.

This study will involve randomizing eligible and consenting women who have been scheduled for labor induction by their obstetrical providers into a pre-hospital cervical ripening (intervention) group or a no pre-hospital ripening (control) group. A trans-cervical Foley balloon (TCFB) will be used for outpatient pre-hospital cervical ripening in women randomized to the intervention group. No pre-hospital ripening will be performed for women in the control group. Both groups will be admitted for induction as scheduled and will undergo labor induction according to a specified, Bishop-score based induction protocol, which may or may not include a TCFB. We will compare the duration of inpatient stays from admission until delivery between the groups as well as satisfaction with the pre-hospital period and labor and delivery experience. Maternal and neonatal outcomes will also be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Intrauterine pregnancy
* Cephalic presentation
* Greater than 36 weeks estimated gestational age
* Reassuring fetal status
* Normal amniotic fluid index
* Clinical indication for induction of labor

Exclusion Criteria:

* Prior cesarean section
* Bishop score on cervical examination ≥ 6
* Unreliable transportation
* Home > 30 minutes from the hospital
* Non-reassuring fetal status
* Abnormal amniotic fluid index
* Other indication for immediate hospitalization

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Salmeen, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Benioff Children's Hospital, San Francisco, California, United States

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Management | Outpatient Transcervical Foley Balloon
Started | 3 | 5
Completed | 0 (Study discontinued prior to data collection.) | 0 (Study discontinued prior to data collection.)
Not Completed | 3 | 5
Not completed — Study discontinued. | 3 | 5

BASELINE CHARACTERISTICS:
Population: Study terminated prior to data collection.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Management | Outpatient Transcervical Foley Balloon | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Duration of Inpatient Time Required to Achieve Delivery
Description: Time from admission to the hospital until delivery
Time Frame: From admission to delivery, expected average of 48 hours
Population: Study terminated prior to data collection.
Arm/Group | Usual Management | Outpatient Transcervical Foley Balloon
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Maternal Satisfaction
Description: Maternal satisfaction with the period leading up to admission and the hospital stay, measured by interview.
Time Frame: up to 48 hours after delivery
Population: Study terminated prior to data collection.
Arm/Group | Usual Management | Outpatient Transcervical Foley Balloon
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Usual Management | Outpatient Transcervical Foley Balloon
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/5
Other Adverse Events (participants affected / at risk) | 0/3 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes